CLINICAL TRIAL: NCT03660943
Title: A Randomized, Double-blind, Placebo-controlled, 2-Injection, 52-Week Study to Evaluate the Efficacy and Safety of Intra-articular Injections of CNTX-4975-05 in Subjects With Chronic, Moderate-to-severe Osteoarthritis Knee Pain
Brief Title: A Clinical Study to Test Efficacy and Safety of Repeat Doses of CNTX-4975-05 in Patients With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNTX-4975i-OA-304
Record Dates: First submitted 2018-08-27; First posted 2018-09-07 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo of 2.0 mL for IA injection
  Interventions: Drug: Placebo
- CNTX-4975-05 (Experimental): Pre-filled glass syringes administered as a single 2.0 mL IA injection
  Interventions: Drug: CNTX-4975-05

INTERVENTIONS:
Drug: Placebo — Receiving Placebo Injection
  Arms: Placebo
Drug: CNTX-4975-05 — Receiving CNTX-4975-05 Injection
  Arms: CNTX-4975-05

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2-injection, 52-week study to evaluate the efficacy and safety of intra-articular injections of CNTX-4975-05 in subjects with chronic, moderate-to-severe osteoarthritis knee pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects between 40 and 95 years of age (inclusive) at the time of the Screening Visit with the ability to comply with answering the electronic diary using the study- provided tablet computers.
* Confirmation of osteoarthritis (OA) of the knee.
* Confirmation of the OA of the index knee.
* Moderate to severe pain in the index knee associated with OA must be stable for a minimum of 6 months prior to Screening, as assessed by the investigator.
* Body Mass Index (BMI) ≤45 kg/m^2
* Must have failed 2 or more prior therapies.

Exclusion Criteria:

* Joint replacement surgery of the index knee at any time, or open surgery of the index knee in the past 24 months.
* Prior arthroscopic surgery of the index knee within 6 months of Screening.
* Any painful conditions of the index knee due to joint disease other than the OA.
* Periarticular pain from any cause.
* Other chronic pain anywhere in the body that requires the use of analgesic medications.
* Instability of the index knee.
* Misalignment (>10 degrees varus or valgus) of the index knee on standing.
* Documented history of neuropathic arthropathy or finding of bony fragmentation in the index knee with imaging.
* Physical/ occupational/ chiropractic therapy for the lower extremities or acupuncture for the lower extremities within 30 days of Screening, or need for such therapy during the study.
* Plans to have surgery, other invasive procedures, or IA injections while participating in the study.
* Has used topical capsaicin on the index knee within 90 days of Screening.
* Current use of opioids for any condition other than for OA of the index knee.
* Corticosteroid injection into the index knee within 90 days of Screening.
* Received IA viscosupplementation (eg, Synvisc®, Hyalgan®) within 90 days of Screening.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (30):
- United States (30):
  - Holland Center for Family Health, Glendale, Arizona
  - GB Family Care, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Med Center Medical Clinic, Carmichael, California
  - TriWest Research Associates, El Cajon, California
  - Arthritis Care and Research Center, Inc. (ACRC Studies), Poway, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Panamerican Health Center, Inc., Miami, Florida
  - Well Pharma Medical Research, Corp, Miami, Florida
  - Quality Research & Medical Center LLC, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Journey Research, Inc., Oldsmar, Florida
  - M&M Clinical Trials Sunrise, Sunrise, Florida
  - Conquest Research, Winter Park, Florida
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Healthcare Research Network, LLC, Flossmoor, Illinois
  - Affinity Clinical Research Institute, Oak Brook, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - BTC of New Bedford, LLC, New Bedford, Massachusetts
  - Healthcare Research Network, Hazelwood, Missouri
  - Office of Robert P. Kaplan, DO, Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - Lillestol Research LLC, Fargo, North Dakota
  - Coastal Carolina Research Center at Arcis Healthcare, LLC dba Lowcountry Orthopaedics & Sports Medicine, North Charleston, South Carolina
  - Heartland Medical, PC, New Tazewell, Tennessee
  - First Surgical Hospital, Bellaire, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - DCT-Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Spectrum Medical, Inc., Danville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- CNTX-4975-05 (Trans-capsaicin): Pre-filled glass syringes administered as a single 2.0 mL IA injection
Period: Overall Study
Arm/Group | Placebo | CNTX-4975-05 (Trans-capsaicin)
Started | 145 | 187
Treated | 140 | 184
Completed | 109 | 134
Not Completed | 36 | 53
Not completed — Adverse Event | 5 | 3
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 7 | 3
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 8 | 15
Not completed — Lack of Efficacy | 9 | 12
Not completed — WITHDRAWAL FOR OTHER TREATMENT; UNABLE TO COMPLETE INJECTION PROCEDURES | 4 | 13

BASELINE CHARACTERISTICS:
Population: The safety population is defined as any subject that received any amount of investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CNTX-4975-05 (Trans-capsaicin) | Total
Number analyzed (Participants) | 140 | 184 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.59) | 62.8 (8.80) | 62.8 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 115 | 199
  Male | 56 | 69 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 56 | 93
  Not Hispanic or Latino | 103 | 128 | 231
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 49 | 86
  White | 97 | 131 | 228
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.40 (5.265) | 32.37 (5.895) | 32.38 (5.623)
Study Baseline WOMAC A (Pain) Domain Score (range 0-50) [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions for knee or hip OA. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).The pain dimension includes 5 items about the amount of pain experienced doing various activities (walking, stair climbing, nocturnal, at rest, weight bearing). The score ranges from 0 to 50. 0 being the best score and 50 being the worst.
  score on a scale | 31.3 (7.2) | 31.6 (7.36) | 31.5 (7.28)
Study Baseline WOMAC B (Stiffness) Domain Score (range 0-20) [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions for knee or hip OA. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).The stiffness dimension includes 2 items about the joint stiffness upon wakening and joint stiffness later in the day. The score ranges from 0 to 20. 0 being the best score and 20 being the worst.
  score on a scale | 13.2 (3.41) | 13.2 (3.15) | 13.2 (3.26)
Study Baseline WOMAC C (Function) Domain Score (range 0-170) [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions for knee or hip OA. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).The physical function dimension asks about the degree of difficulty in doing 17 activities due to the reference joint. The score ranges from 0 to 170. 0 being the best score and 170 being the worst.
  score on a scale | 107.9 (26.71) | 109.5 (25.89) | 108.8 (26.22)
Average Weekly Pain with Walking NPRS (0-10) Score [Mean (Standard Deviation); unit: score on a scale] — Average daily OA pain in the index knee while walking was evaluated using a 0 to 10 Numerical Pain Rating Scale (NPRS) (0 = no pain and 10 = worst possible pain). 0 was the best score and 10 was the worst score.
  score on a scale | 6.933 (1.021) | 7.013 (0.9950) | 6.978 (1.0055)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in WOMAC A (Pain) Dimension
Description: The Western Ontario and McMaster Universities developed the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score to use among patients with knee and/or hip OA. The WOMAC is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).
  The WOMAC is a self-administered index that contains 24 items asked in relation to the index knee joint. The WOMAC has 3 dimensions: Pain (Subscale A), Stiffness (Subscale B), and Physical Function (Subscale C). Lower scores mean a better outcome and higher scores mean a worse outcome.
  The pain dimension includes 5 items about the amount of pain experienced doing various activities (walking, stair climbing, nocturnal, at rest, weight bearing). The score ranges from 0 to 50.
Time Frame: Baseline, Week 12
Population: The intent to treat (ITT) population included all randomized subjects who received any amount of investigational product and all observed data
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 125 | 164
score on a scale | -14.13 (12.217) | -17.16 (12.266)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; The MMRM analysis included the change from study baseline in scores as the dependent variable, with terms for treatment, pooled study center, study baseline K-L grade category for the index knee, study baseline BMI category, study baseline OA type (unilateral or bilateral knee OA), sex, study visit, treatment by visit interaction, and study baseline score as covariates, using an unstructured covariance structure; Test type: Superiority; p = 0.0833, Mixed Models Analysis; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-4.42 to 0.27], Standard Error of Mean 1.192

2. Secondary Outcome: Change From Baseline in Average Weekly Pain With Walking (NPRS 0-10) in the Index Knee
Description: Average daily OA pain in the index knee while walking was evaluated using a 0 to 10 Numerical Pain Rating Scale (NPRS) (0 = no pain and 10 = worst possible pain). 0 was the best score and 10 was the worst score.
  Subjects used an ePRO at bedtime (9:00 PM ± 3 hours) to record on a daily basis their average daily OA knee pain score with walking during the previous 24 hours.
Time Frame: Baseline, Week 12
Population: The intent to treat (ITT) population included all randomized subjects who received any amount of investigational product and all observed data as collected in the daily diary
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 128 | 170
score on a scale | -2.99 (0.213) | -3.41 (0.197)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The number of NPRS subjects differed from the WOMAC outcomes because of differences in missing data; p = 0.0935, Mixed Models Analysis; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.91 to 0.07], Standard Error of Mean 0.251

3. Secondary Outcome: Mean Change From Study Baseline in WOMAC B (Stiffness) Dimension
Description: The Western Ontario and McMaster Universities developed the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score to use among patients with knee and/or hip OA. The WOMAC is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).
  The WOMAC is a self-administered index that contains 24 items asked in relation to the index knee joint. The WOMAC has 3 dimensions: Pain (Subscale A), Stiffness (Subscale B), and Physical Function (Subscale C). Lower scores mean a better outcome and higher scores mean a worse outcome.
  The stiffness dimension has 2 items: joint stiffness upon wakening and joint stiffness later in the day. The score ranges from 0 to 20.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 125 | 164
score on a scale | -5.36 (0.434) | -6.58 (0.404)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0163, Mixed Models Analysis; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.22 to -0.23], Standard Error of Mean 0.506

4. Secondary Outcome: Mean Change From Study Baseline in WOMAC C (Function) Dimension
Description: The Western Ontario and McMaster Universities developed the Western Ontario and McMaster Universities Arthritis Index (WOMAC) score to use among patients with knee and/or hip OA. The WOMAC is a validated, multidimensional measure of pain, stiffness, and physical functional disability that is sensitive to the effects of drugs or other interventions. This study used the 11-box NPRS format ranging from 0 (none or no pain/stiffness/difficulty) to 10 (extreme).
  The WOMAC is a self-administered index that contains 24 items asked in relation to the index knee joint. The WOMAC has 3 dimensions: Pain (Subscale A), Stiffness (Subscale B), and Physical Function (Subscale C). Lower scores mean a better outcome and higher scores mean a worse outcome.
  The function dimension asks about the degree of difficulty in doing 17 activities due to the reference joint. The score ranges from 0 to 170.
Time Frame: Baseline, Week12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | CNTX-4975-05
Number analyzed (Participants) | 125 | 164
score on a scale | -49.03 (3.541) | -57.02 (3.307)
Statistical Analysis 1: Comparison: Placebo vs CNTX-4975-05; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0509, Mixed Models Analysis; Mean Difference (Final Values) = -7.99, 95% CI 2-sided [-16.01 to 0.03], Standard Error of Mean 4.076

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Placebo | CNTX-4975-05 (Trans-capsaicin)
All-Cause Mortality (participants affected / at risk) | 0/140 | 2/184
Serious Adverse Events (participants affected / at risk) | 9/140 | 9/184
Other Adverse Events (participants affected / at risk) | 34/140 | 70/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | CNTX-4975-05 (Trans-capsaicin) (N=184)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Peritoneal bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | CNTX-4975-05 (Trans-capsaicin) (N=184)
Viral upper respiratory tract infection (Infections and infestations) | 5 | 13
Upper respiratory tract infection (Infections and infestations) | 6 | 4
Bronchitis (Infections and infestations) | 2 | 6
Sinusitis (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 7
Headache (Nervous system disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 1 | 5
Anaemia (Blood and lymphatic system disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03660943/Prot_SAP_000.pdf